CLINICAL TRIAL: NCT01677858
Title: A Phase 1/2 Study of Weekly Carfilzomib in Combination With Dexamethasone for Progressive Multiple Myeloma
Brief Title: A Study of Weekly Carfilzomib in Combination With Dexamethasone for Progressive Multiple Myeloma
Acronym: CHAMPION 1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2012-002; 20130403 (Other: Amgen Inc.)
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carfilzomib (Experimental): In phase 1 participants were assigned to one of four sequential dose-escalating cohorts to receive 45, 56, 70 or 88 mg/m² carfilzomib administered by intravenous (IV) infusion on days 1, 8 and 15 of each 28-day cycle. Participants also received 40 mg dexamethasone IV or orally on days 1, 8, 15 and 22 for the first 8 cycles; starting with cycle 9, dexamethasone was administered only on days 1, 8, and 15.
  In phase 2 participants received carfilzomib at the maximum tolerated dose (MTD) established in the Phase 1 portion of the study on days 1, 8 and 15 plus 40 mg dexamethasone IV or orally at the same schedule as used in the Phase 1 portion of the study.
  Participants were treated until confirmed progressive disease, unacceptable toxicity, withdrew consent for further treatment, were lost to follow-up, died, or the sponsor closed the study.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib was administered as a 30-minute IV infusion on days 1, 8, and 15 of each 28-day treatment cycle.
  Other Names: Krypolis
Drug: Dexamethasone — Dexamethasone was administered at a dose of 40 mg IV or orally (PO) on days 1, 8, 15, and 22 for the first 8 cycles; starting with cycle 9 dexamethasone was administered on days 1, 8, and 15.

SUMMARY:
The study had the following primary objectives:

* Phase 1: to determine the maximum tolerated dose (MTD) of once-weekly (QW) carfilzomib and dexamethasone for patients with relapsed or refractory multiple myeloma who have received 1 to 3 prior therapies
* Phase 2: to estimate the overall response rate (ORR) for patients with relapsed or refractory multiple myeloma who received 1 to 3 prior therapies treated with carfilzomib and dexamethasone QW at the MTD established in phase 1.

DETAILED DESCRIPTION:
This is a Phase 1/2, multicenter, single-arm, nonrandomized, open-label and dose-escalation study of weekly carfilzomib and dexamethasone for patients with progressive multiple myeloma. The Phase 1 dose escalation portion will enroll patients into sequential dose-escalating cohorts consisting of 3 patients each to establish the maximum tolerated dose (MTD) of carfilzomib administered weekly as a 30 minute intravenous (IV) infusion with dexamethasone. The Phase 2 portion will enroll patients using the MTD established for carfilzomib from the Phase 1 portion of the study. Dexamethasone will be administered IV or orally at the same dose and schedule as used in the Phase 1 portion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Multiple myeloma with relapsing or progressive disease at study entry
2. Measurable disease, as defined by 1 or more of the following (assessed within 21 days prior to enrollment):

   1. Serum M-protein ≥ 0.5 g/dL, or
   2. Urine M-protein ≥ 200 mg/24 hours, or
   3. Only in patients who do not meet a or b, then use serum free light chain (SFLC) > 100 mg/L (involved light chain) and an abnormal kappa/lambda ratio
3. Prior treatment with 1 to 3 prior regimens for multiple myeloma for Phase 1 and Phase 2 (induction therapy followed by stem cell transplant and consolidation/maintenance therapy will be considered as 1 line of therapy
4. Age ≥ 18 years
5. Life expectancy ≥ 6 months
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
7. Adequate hepatic function within 21 days prior to enrollment, with bilirubin < 1.5 × the upper limit of normal (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 × ULN
8. Left ventricular ejection fraction (LVEF) ≥ 40%. 2-D transthoracic echocardiogram (ECHO) is the preferred method of evaluation. Multigated acquisition scan (MUGA) is acceptable if ECHO is not available
9. Absolute neutrophil count (ANC) ≥ 1000/mm³ within 21 days prior to enrollment. Screening ANC is to be independent of growth factor support for ≥ 1 week
10. Hemoglobin ≥ 8.0 g/dL within 21 days prior to enrollment. Use of erythropoietic stimulating factors and red blood cell (RBC) transfusions per institutional guidelines is allowed; however, most recent RBC transfusion must have been at least 7 days prior to obtaining screening hemoglobin
11. Platelet count ≥ 50,000/mm³ (≥ 30,000/mm³ if myeloma involvement in the bone marrow is > 50%) within 21 days prior to enrollment. Patients must not have received platelet transfusions for at least 7 days prior to obtaining the screening platelet count
12. Calculated or measured creatinine clearance (CrCl) of ≥ 30 mL/min within 21 days prior to enrollment. Calculation based on standard formula, such as the Cockcroft and Gault: [(140 - Age) x Mass (kg) / (72 x Creatinine mg/dL)]; multiply result by 0.85 if female
13. Written informed consent in accordance with federal, local, and institutional guidelines
14. Female patients of childbearing potential (FCBP) must have a negative serum pregnancy test within 21 days prior to enrollment and agree to use an effective method of contraception during and for 3 months following last dose of drug (more frequent pregnancy tests may be conducted if required per local regulations). Postmenopausal females (> 45 years old and without menses for > 1 year) and surgically sterilized females are exempt from a pregnancy test
15. Male patients must agree to use an effective barrier method of contraception during study and for 3 months following the last dose if sexually active with an FCBP

Exclusion Criteria:

1. Multiple myeloma of Immunoglobulin M (IgM) subtype
2. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
3. Plasma cell leukemia (> 2.0 × 10^9/L circulating plasma cells by standard differential)
4. Waldenström's macroglobulinemia
5. Amyloidosis
6. Glucocorticoid therapy (prednisone > 30 mg/day or equivalent) within 7 days prior to enrollment
7. Cytotoxic chemotherapy with approved or investigational anticancer therapeutics within 28 days prior to enrollment
8. Treatment with bortezomib (Velcade®), thalidomide (Thalomid®) or lenalidomide (Revlimid®) within 21 days prior to enrollment
9. Focal radiation therapy within 7 days prior to enrollment. Radiation therapy to an extended field involving a significant volume of bone marrow within 21 days prior to enrollment (ie, prior radiation must have been to < 30% of the bone marrow)
10. Immunotherapy within 21 days prior to enrollment
11. Major surgery within 21 days prior to enrollment
12. Active congestive heart failure (New York Heart Association [NYHA] Classes III to IV), symptomatic ischemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within 6 months prior to enrollment
13. Acute active infection requiring systemic antibiotics, antiviral (except antiviral therapy directed at hepatitis B virus [HBV]), or antifungal agents within 14 days prior to enrollment
14. Known human immunodeficiency virus (HIV) seropositivity
15. Known hepatitis B or C virus infection (except for patients with HBV who are receiving and responding to HBV antiviral therapy: these patients are allowed)
16. Patients with known cirrhosis
17. Second malignancy within the past 3 years, except:

    1. Adequately treated basal cell or squamous cell skin cancer
    2. Carcinoma in situ of the cervix
    3. Prostate cancer < Gleason score 6 with stable prostate-specific antigen (PSA) over 12 months
    4. Breast carcinoma in situ with full surgical resection
    5. Treated medullary or papillary thyroid cancer
18. Patients with myelodysplastic syndrome
19. Significant neuropathy (Grades 3 to 4) within 14 days prior to enrollment
20. Female patients who are pregnant or lactating
21. Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib)
22. Prior carfilzomib treatment
23. Prior participation in any Onyx-sponsored Phase 3 trial
24. Patients with contraindication to dexamethasone
25. Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment
26. Ongoing graft-versus-host disease
27. Patients with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to enrollment
28. Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to enrollment
29. Any other clinically significant medical disease or psychiatric condition that, in the Investigator's opinion, may interfere with protocol adherence or a patient's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2012-07-04; Primary Completion 2016-07-22 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (35):
- United States (35):
  - Arizona Oncology Associates, Tucson, Arizona
  - Comprehensive Blood and Cancer Center (CCBC), Bakersfield, California
  - California Cancer Associates for Research and Excellence, Encinitas, California
  - Robert A. Moss, M.D., FACP, Inc., Fountain Valley, California
  - California Cancer Associates for Research and Excellence, Fresno, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Monterey Bay Oncology, Salinas, California
  - Sansum Clinic, Santa Barbara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - James R. Berenson M.D. Inc., West Hollywood, California
  - The Oncology Insititute of Hope and Innovation, Whittier, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Florida Cancer Specialists - North, Tampa, Florida
  - Illinois Cancer Care, Galesburg, Illinois
  - Illinois Cancer Specialists, Hinsdale, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Fort Wayne Oncology & Hematology, Fort Wayne, Indiana
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - Center for Cancer and Blood Disorders (CCBD), Bethesda, Maryland
  - Hematology-Oncology Associates of Northern NJ, PA, Morristown, New Jersey
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Clinical Research Alliance, New York, New York
  - Hudson Valley Hematology Oncology Associates, Poughkeepsie, New York
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Tennessee Oncology, PLLC, Chattanooga, Tennessee
  - St. Joseph Regional Cancer Center, Bryan, Texas
  - Millennium Oncology, Houston, Texas
  - Waldron Medical Research and Development Center, Houston, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Center at Cancer Therapy & Research Center at The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Blood and Cancer Center of East Texas, Tyler, Texas
  - Shenandoah Oncology, PC, Winchester, Virginia
  - Northwest Cancer Specialists, Vancouver, Washington
  - Yakima Valley Memorial Hospital/ North Star Lodge, Yakima, Washington

REFERENCES:
- [Background] Moreau P, Stewart KA, Dimopoulos M, Siegel D, Facon T, Berenson J, Raje N, Berdeja JG, Orlowski RZ, Yang H, Ma H, Klippel Z, Zahlten-Kumeli A, Mezzi K, Iskander K, Mateos MV. Once-weekly (70 mg/m2 ) vs twice-weekly (56 mg/m2 ) dosing of carfilzomib in patients with relapsed or refractory multiple myeloma: A post hoc analysis of the ENDEAVOR, A.R.R.O.W., and CHAMPION-1 trials. Cancer Med. 2020 May;9(9):2989-2996. doi: 10.1002/cam4.2945. Epub 2020 Feb 28. PMID 32108443
- [Derived] Berenson JR, Cartmell A, Bessudo A, Lyons RM, Harb W, Tzachanis D, Agajanian R, Boccia R, Coleman M, Moss RA, Rifkin RM, Patel P, Dixon S, Ou Y, Anderl J, Aggarwal S, Berdeja JG. CHAMPION-1: a phase 1/2 study of once-weekly carfilzomib and dexamethasone for relapsed or refractory multiple myeloma. Blood. 2016 Jun 30;127(26):3360-8. doi: 10.1182/blood-2015-11-683854. Epub 2016 May 12. PMID 27207788

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 32 centers in the United States. Participants were enrolled from September 2012 to September 2014.
Pre-assignment Details: In phase 1 participants were enrolled into 1 of 4 sequential dose-escalating cohorts to establish the maximum tolerated dose (MTD) of carfilzomib plus dexamethasone. In phase 2 participants were enrolled to evaluate the efficacy and safety of carfilzomib plus dexamethasone at the MTD established in phase 1.
Groups:
- Phase 1: Carfilzomib 45 mg/m²: Participants received carfilzomib administered by intravenous (IV) infusion on days 1, 8 and 15 of each 28-day cycle. The carfilzomib dose was 20 mg/m² on day 1 of cycle 1; thereafter, subsequent carfilzomib dosing was 45 mg/m². Participants also received 40 mg dexamethasone IV or orally on days 1, 8, 15 and 22 for the first 8 cycles; starting with cycle 9, dexamethasone was administered only on days 1, 8, and 15.
- Phase 1: Carfilzomib 56 mg/m²: Participants received carfilzomib administered by intravenous (IV) infusion on days 1, 8 and 15 of each 28-day cycle. The carfilzomib dose was 20 mg/m² on day 1 of cycle 1; thereafter, subsequent carfilzomib dosing was 56 mg/m². Participants also received 40 mg dexamethasone IV or orally on days 1, 8, 15 and 22 for the first 8 cycles; starting with cycle 9, dexamethasone was administered only on days 1, 8, and 15.
- Phase 1: Carfilzomib 70 mg/m²; Phase 2: Carfilzomib 70 mg/m²: Participants received carfilzomib administered by intravenous (IV) infusion on days 1, 8 and 15 of each 28-day cycle. The carfilzomib dose was 20 mg/m² on day 1 of cycle 1; thereafter, subsequent carfilzomib dosing was 70 mg/m². Participants also received 40 mg dexamethasone IV or orally on days 1, 8, 15 and 22 for the first 8 cycles; starting with cycle 9, dexamethasone was administered only on days 1, 8, and 15.
- Phase 1: Carfilzomib 88 mg/m²: Participants received carfilzomib administered by intravenous (IV) infusion on days 1, 8 and 15 of each 28-day cycle. The carfilzomib dose was 20 mg/m² on day 1 of cycle 1; thereafter, subsequent carfilzomib dosing was 88 mg/m². Participants also received 40 mg dexamethasone IV or orally on days 1, 8, 15 and 22 for the first 8 cycles; starting with cycle 9, dexamethasone was administered only on days 1, 8, and 15.
Period: Overall Study
Arm/Group | Phase 1: Carfilzomib 45 mg/m² | Phase 1: Carfilzomib 56 mg/m² | Phase 1: Carfilzomib 70 mg/m² | Phase 1: Carfilzomib 88 mg/m² | Phase 2: Carfilzomib 70 mg/m²
Started | 3 | 3 | 15 | 6 | 89
Completed | 0 (Completed indicates participants ongoing in study) | 1 (Completed indicates participants ongoing in study) | 1 (Completed indicates participants ongoing in study) | 0 (Completed indicates participants ongoing in study) | 4 (Completed indicates participants ongoing in study)
Not Completed | 3 | 2 | 14 | 6 | 85
Not completed — Adverse Event | 0 | 0 | 2 | 3 | 13
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 2 | 0 | 12
Not completed — Progressive Disease | 2 | 1 | 9 | 3 | 43
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 15
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Carfilzomib 45 mg/m² | Phase 1: Carfilzomib 56 mg/m² | Phase 1: Carfilzomib 70 mg/m² | Phase 1: Carfilzomib 88 mg/m² | Phase 2: Carfilzomib 70 mg/m² | Total
Number analyzed (Participants) | 3 | 3 | 15 | 6 | 89 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (15.6) | 73.7 (2.1) | 62.4 (10.4) | 58.2 (8.8) | 68.7 (9.6) | 67.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 5 | 40 | 52
  Male | 2 | 1 | 11 | 1 | 49 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 10 | 11
  Not Hispanic or Latino | 3 | 3 | 15 | 5 | 79 | 105
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 2 | 11 | 6 | 79 | 101
  Black or African American | 0 | 1 | 2 | 0 | 6 | 9
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  American Indian or Alaskan Native | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Other | 0 | 0 | 2 | 0 | 1 | 3
  Unknown | 0 | 0 | 0 | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a participants disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active; 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, no self-care, confined to bed or chair; 5 = Dead.
  Participants
    0 (Fully active) | 1 | 2 | 6 | 3 | 39 | 51
    1 (Restrictive but ambulatory) | 2 | 1 | 9 | 3 | 50 | 65

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: The MTD was defined as the highest carfilzomib dose at which < 33% of participants had a treatment-related DLT during the first 28-day cycle. A DLT was categorized as nonhematologic or hematologic and defined as follows:
  Nonhematologic:
  * ≥ grade 3 nonhematological toxicity (excluding nausea, vomiting, diarrhea, fatigue lasting < 14 days, increased serum creatinine or electrolyte abnormalities not clinically significant or requiring treatment)
  * ≥ grade 3 acute kidney injury (creatinine > 3 x baseline or > 4.0 mg/dL) lasting > 72 hours
  * ≥ grade 3 nausea, vomiting, or diarrhea uncontrolled by maximal antiemetic/antidiarrheal therapy
  Hematologic:
  * grade 4 neutropenia (absolute neutrophil count [ANC] < 500/mm³) for > 7 days
  * febrile neutropenia (ANC < 1000/mm³ with a fever ≥ 38.3ºC) of any duration
  * grade 4 thrombocytopenia (< 25 000/mm³) for > 14 days, despite holding treatment
  * grade 3 or 4 thrombocytopenia (< lower limit of normal) associated with > grade 1 bleeding
Time Frame: 28 days
Population: Participants in phase 1 who received at least 1 dose of any investigational product (carfilzomib or dexamethasone).
Measure: Number; unit: participants
Groups:
- Phase 1 Carfilzomib 45 mg/m²: Participants received carfilzomib administered by intravenous (IV) infusion on days 1, 8 and 15 of each 28-day cycle. The carfilzomib dose was 20 mg/m² on day 1 of cycle 1; thereafter, subsequent carfilzomib dosing was 45 mg/m². Participants also received 40 mg dexamethasone IV or orally on days 1, 8, 15 and 22 for the first 8 cycles; starting with cycle 9, dexamethasone was administered only on days 1, 8, and 15.
Arm/Group | Phase 1 Carfilzomib 45 mg/m² | Phase 1: Carfilzomib 56 mg/m² | Phase 1: Carfilzomib 70 mg/m² | Phase 1: Carfilzomib 88 mg/m²
Number analyzed (Participants) | 3 | 3 | 15 | 6
participants | 0 | 0 | 1 | 2
Statistical Analysis 1: Comparison: Phase 1 Carfilzomib 45 mg/m² vs Phase 1: Carfilzomib 56 mg/m² vs Phase 1: Carfilzomib 70 mg/m² vs Phase 1: Carfilzomib 88 mg/m²; Test type: Other; Maximum Tolerated Dose (mg/m²) = 70

2. Primary Outcome: Overall Response Rate (ORR)
Description: Disease response was evaluated by the investigator according to the International Myeloma Working Group Uniform Response Criteria (IMWG-URC). ORR was defined as the percentage of participants with a best overall response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR).
  sCR: As for CR, normal serum free light chain (SFLC) ratio and no clonal cells in bone marrow (BM).
  CR: No immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas and < 5% plasma cells in BM.
  VGPR: Serum and urine M-protein detectable by immunofixation but not electrophoresis or ≥ 90% reduction in serum M-protein with urine M-protein <100 mg/24 hours. A ≥ 50% reduction in the size of soft tissue plasmacytomas if present at baseline.
  PR: ≥ 50% reduction of serum M-protein and reduction in urine M-protein by ≥ 90% or to < 200 mg/24 hours. A ≥ 50% reduction in the size of soft tissue plasmacytomas if present at baseline.
Time Frame: Disease response was assessed once every treatment cycle (28 days) and 30 days after last dose; the median overall treatment duration was 33.6 weeks.
Population: Participants who received at least 1 dose of any investigational product (carfilzomib or dexamethasone).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1+2: Carfilzomib 70 mg/m²: Participants received carfilzomib administered by intravenous (IV) infusion on days 1, 8 and 15 of each 28-day cycle. The carfilzomib dose was 20 mg/m² on day 1 of cycle 1; thereafter, subsequent carfilzomib dosing was 70 mg/m². Participants also received 40 mg dexamethasone IV or orally on days 1, 8, 15 and 22 for the first 8 cycles; starting with cycle 9, dexamethasone was administered only on days 1, 8, and 15.
Arm/Group | Phase 1: Carfilzomib 45 mg/m² | Phase 1: Carfilzomib 56 mg/m² | Phase 1: Carfilzomib 70 mg/m² | Phase 1: Carfilzomib 88 mg/m² | Phase 2: Carfilzomib 70 mg/m² | Phase 1+2: Carfilzomib 70 mg/m²
Number analyzed (Participants) | 3 | 3 | 15 | 6 | 89 | 104
percentage of participants | 33.3 [0.8 to 90.6] | 100 [29.2 to 100.0] | 93.3 [68.1 to 99.8] | 66.7 [22.3 to 95.7] | 74.2 [63.8 to 82.9] | 76.9 [67.6 to 84.6]

3. Secondary Outcome: Clinical Benefit Response Rate
Description: Clinical benefit rate was defined as the percentage of participants whose best response was sCR, CR, VGPR, PR, or minimal response (MR), where MR is defined by the European Group for Blood and Marrow Transplant (EBMT) criteria as a 25% to 49% reduction in the level of serum M-protein or a 50% to 89% reduction in 24-hour urinary M-protein, which still exceeds 200 mg /24 hour, maintained for a minimum of 8 weeks.
Time Frame: as for outcome 2
Population: Participants who received at least 1 dose of any investigational product (carfilzomib or dexamethasone).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Carfilzomib 45 mg/m² | Phase 1: Carfilzomib 56 mg/m² | Phase 1: Carfilzomib 70 mg/m² | Phase 1: Carfilzomib 88 mg/m² | Phase 2: Carfilzomib 70 mg/m² | Phase 1+2: Carfilzomib 70 mg/m²
Number analyzed (Participants) | 3 | 3 | 15 | 6 | 89 | 104
percentage of participants | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0] | 100.0 [78.2 to 100.0] | 83.3 [35.9 to 99.6] | 80.9 [71.2 to 88.5] | 83.7 [75.1 to 90.2]

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time from first dose to the earlier of disease progression or death due to any cause. The duration of PFS was calculated using Kaplan-Meier methods; participants with no baseline and/or post-baseline disease assessments, who started a new anticancer therapy before documentation of disease progression or death, died or had disease progression immediately after more than 1 consecutively missed disease assessment visit or who were alive without documentation of disease progression before the data cutoff date were censored.
  Participants were evaluated for disease response and progression by the investigator according to the IMWG-URC.
Time Frame: From randomization until the data cut-off date of 22 July 2016; median follow-up time for PFS was 13.8 months
Population: Participants who received at least 1 dose of any investigational product (carfilzomib or dexamethasone).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: Carfilzomib 45 mg/m² | Phase 1: Carfilzomib 56 mg/m² | Phase 1: Carfilzomib 70 mg/m² | Phase 1: Carfilzomib 88 mg/m² | Phase 2: Carfilzomib 70 mg/m² | Phase 1+2: Carfilzomib 70 mg/m²
Number analyzed (Participants) | 3 | 3 | 15 | 6 | 89 | 104
months | 13.6 [6.4 to 20.7] | NA [41.7 to NA] — Could not be estimated due to the low number of events | 21.0 [4.2 to NA] — Could not be estimated due to the low number of events | 12.9 [3.9 to 20.0] | 15.3 [10.0 to 20.2] | 16.2 [10.2 to 21.0]

5. Secondary Outcome: Time To Progression
Description: Time to progression (TTP) was defined as the time from first dose to disease progression evaluated by the investigator according to the International Myeloma Working Group Uniform Response Criteria (IMWG-URC). TTP was calculated using Kaplan-Meier methods; participants with no baseline and/or post-baseline disease assessments, who started a new anticancer therapy before documentation of disease progression or death, died or had disease progression immediately after more than 1 consecutively missed disease assessment visit or who were alive without documentation of disease progression before the data cutoff date were censored.
Time Frame: From randomization until the data cut-off date of 22 July 2016; median follow-up time for TTP was 13.4 months
Population: Participants who received at least 1 dose of any investigational product (carfilzomib or dexamethasone).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: Carfilzomib 45 mg/m² | Phase 1: Carfilzomib 56 mg/m² | Phase 1: Carfilzomib 70 mg/m² | Phase 1: Carfilzomib 88 mg/m² | Phase 2: Carfilzomib 70 mg/m² | Phase 1+2: Carfilzomib 70 mg/m²
Number analyzed (Participants) | 3 | 3 | 15 | 6 | 89 | 104
months | 13.6 [6.4 to 20.7] | NA [41.7 to NA] — Could not be estimated due to the low number of events | 21.0 [4.2 to NA] — Could not be estimated due to the low number of events | 12.9 [3.9 to 20.0] | 16.2 [10.2 to 20.2] | 17.2 [10.6 to 21.7]

6. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) was defined as the time from first evidence of PR or better to disease progression or death due to any cause. DOR was calculated using Kaplan-Meier methods; Participants with no baseline disease assessments, starting a new anticancer therapy before documentation of disease progression or death, death or disease progression immediately after more than 1 consecutively missed disease assessment visit, or alive without documentation of disease progression before the data cut-off date were censored.
Time Frame: From randomization until the data cut-off date of 22 July 2016; median follow-up time for DOR was 14.3 months
Population: Participants who received at least 1 dose of any investigational product (carfilzomib or dexamethasone) with a best overall response of sCR, CR, VGPR, or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: Carfilzomib 45 mg/m² | Phase 1: Carfilzomib 56 mg/m² | Phase 1: Carfilzomib 70 mg/m² | Phase 1: Carfilzomib 88 mg/m² | Phase 2: Carfilzomib 70 mg/m² | Phase 1+2: Carfilzomib 70 mg/m²
Number analyzed (Participants) | 1 | 3 | 14 | 4 | 66 | 80
months | 18.9 [NA to NA] — Could not be estimated due to the low number of events | NA [39.9 to NA] — Could not be estimated due to the low number of events | 16.3 [3.3 to NA] — Could not be estimated due to the low number of events | 11.9 [11.1 to 18.9] | 18.0 [13.7 to 21.9] | 18.0 [14.5 to 21.9]

7. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events were graded using National Cancer Institute-Common Terminology Criteria for Adverse Events (version 4.03).
Time Frame: From the first day of study treatment and within 30 days of the last day of study treatment; median duration of treatment was 33.6 weeks.
Population: Participants who received at least 1 dose of any investigational product (carfilzomib or dexamethasone).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Carfilzomib 45 mg/m² | Phase 1: Carfilzomib 56 mg/m² | Phase 1: Carfilzomib 70 mg/m² | Phase 1: Carfilzomib 88 mg/m² | Phase 2: Carfilzomib 70 mg/m²
Number analyzed (Participants) | 3 | 3 | 15 | 6 | 89
Participants
  All adverse events | 3 | 3 | 15 | 6 | 89
  Adverse events ≥ grade 3 | 1 | 2 | 9 | 5 | 60
  Serious adverse events | 1 | 0 | 4 | 1 | 35
  AE leading to discontinuation of carfilzomib & dex | 0 | 0 | 2 | 3 | 14
  AE leading to discontinuation of carfilzomib | 0 | 0 | 2 | 3 | 14
  Fatal adverse events | 0 | 0 | 0 | 0 | 5

8. Secondary Outcome: Time to Maximum Plasma Concentration of Carfilzomib
Time Frame: Day 1 cycle 1 (20 mg/m² carfilzomib), cycle 1 day 15 (phase 1 70 and 88 mg/m² carfilzomib), and cycle 2 day 15 (phase 2 70 mg/m² carfilzomib) from predose to 4 hours after the end of the infusion.
Population: Pharmacokinetic (PK) analyses were conducted for participants assigned to cohorts 3 and 4 in phase 1 (70 and 88 mg/m² carfilzomib) and a subset of participants in phase 2; only participants for whom PK parameters could be calculated were included in the analyses.
Measure: Median (Full Range); unit: hours
Groups:
- Carfilzomib 20 mg/m²: Participants in phase 1 and phase 2 received carfilzomib 20 mg/m² administered by intravenous (IV) infusion on day 1 cycle 1.
- Carfilzomib 70 mg/m²: Participants in phase 1 and phase 2 received carfilzomib 70 mg/m² administered by intravenous (IV) infusion from day 8 cycle 1 onwards.
- Carfilzomib 88 mg/m²: Participants in phase 1 received carfilzomib 88 mg/m² administered by intravenous (IV) infusion from day 8 cycle 1 onwards.
Arm/Group | Carfilzomib 20 mg/m² | Carfilzomib 70 mg/m² | Carfilzomib 88 mg/m²
Number analyzed (Participants) | 26 | 21 | 5
hours | 0.25 [0.17 to 0.75] | 0.25 [0.08 to 0.58] | 0.25 [0.25 to 0.58]

9. Secondary Outcome: Maximum Plasma Concentration of Carfilzomib
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Carfilzomib 20 mg/m² | Carfilzomib 70 mg/m² | Carfilzomib 88 mg/m²
Number analyzed (Participants) | 26 | 21 | 5
ng/mL | 789 (65.5) | 2390 (30.7) | 3090 (27.3)

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of Last Quantifiable Concentration (AUClast) for Carfilzomib
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Carfilzomib 20 mg/m² | Carfilzomib 70 mg/m² | Carfilzomib 88 mg/m²
Number analyzed (Participants) | 26 | 21 | 5
hr*ng/mL | 281 (52.7) | 1040 (21.7) | 1210 (31.4)

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUCinf) fo Carfilzomib
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Carfilzomib 20 mg/m² | Carfilzomib 70 mg/m² | Carfilzomib 88 mg/m²
Number analyzed (Participants) | 25 | 16 | 4
hr*ng/mL | 259 (28.0) | 1040 (21.6) | 1160 (34.8)

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve During the Dosing Interval (0-168 Hours) for Carfilzomib
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Carfilzomib 20 mg/m² | Carfilzomib 70 mg/m² | Carfilzomib 88 mg/m²
Number analyzed (Participants) | 25 | 16 | 4
hr*ng/mL | 259 (28.0) | 1040 (21.6) | 1160 (34.8)

13. Secondary Outcome: Volume of Distribution Observed at Steady State (Vss) for Carfilzomib
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Carfilzomib 20 mg/m² | Carfilzomib 70 mg/m² | Carfilzomib 88 mg/m²
Number analyzed (Participants) | 24 | 16 | 4
liters | 17.0 (133.3) | 14.2 (54.2) | 7.87 (78.4)

14. Secondary Outcome: Terminal Half-life (T1/2,z) for Carfilzomib
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Carfilzomib 20 mg/m² | Carfilzomib 70 mg/m² | Carfilzomib 88 mg/m²
Number analyzed (Participants) | 25 | 15 | 4
hours | 0.648 (49) | 0.883 (24.6) | 0.816 (17.1)

15. Secondary Outcome: Clearance of Carfilzomib After IV Infusion
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters/hour
Arm/Group | Carfilzomib 20 mg/m² | Carfilzomib 70 mg/m² | Carfilzomib 88 mg/m²
Number analyzed (Participants) | 25 | 16 | 4
liters/hour | 147 (31.0) | 131 (29.6) | 138 (35.0)

16. Secondary Outcome: Mean Residence Time Observed From Time Zero to Infinity (MRT0-∞) for Carfilzomib
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Carfilzomib 20 mg/m² | Carfilzomib 70 mg/m² | Carfilzomib 88 mg/m²
Number analyzed (Participants) | 24 | 16 | 4
hours | 0.118 (130.5) | 0.108 (55.4) | 0.0571 (110.0)

ADVERSE EVENTS:
Time Frame: From the first day of study treatment and within 30 days of the last day of study treatment; median duration of treatment was 33.6 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Phase 1: Carfilzomib 45 mg/m² | Phase 1: Carfilzomib 56 mg/m² | Phase 1: Carfilzomib 70 mg/m² | Phase 1: Carfilzomib 88 mg/m² | Phase 2: Carfilzomib 70 mg/m²
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 4/15 | 1/6 | 35/89
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 15/15 | 6/6 | 87/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Carfilzomib 45 mg/m² (N=3) | Phase 1: Carfilzomib 56 mg/m² (N=3) | Phase 1: Carfilzomib 70 mg/m² (N=15) | Phase 1: Carfilzomib 88 mg/m² (N=6) | Phase 2: Carfilzomib 70 mg/m² (N=89)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 2
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 2
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 4
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 5
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Haematuria traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 6
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Carfilzomib 45 mg/m² (N=3) | Phase 1: Carfilzomib 56 mg/m² (N=3) | Phase 1: Carfilzomib 70 mg/m² (N=15) | Phase 1: Carfilzomib 88 mg/m² (N=6) | Phase 2: Carfilzomib 70 mg/m² (N=89)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 5 | 1 | 25
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1 | 22
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 4
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 5
Porokeratosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Amblyopia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Blindness (Eye disorders) | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 1 | 2
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 1
Dry eye (Eye disorders) | 0 | 1 | 1 | 1 | 1
Eye discharge (Eye disorders) | 0 | 1 | 1 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 2 | 1 | 2 | 5
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 4
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 8
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 6 | 1 | 11
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 9 | 2 | 26
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 5
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2
Gastrointestinal tract irritation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 3
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Loose tooth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 7 | 3 | 36
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3
Tooth loss (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 4 | 2 | 13
Asthenia (General disorders) | 0 | 1 | 4 | 0 | 9
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 3
Chills (General disorders) | 0 | 1 | 4 | 0 | 5
Cyst (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 2 | 9 | 3 | 47
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 2 | 0 | 3
Infusion site extravasation (General disorders) | 0 | 0 | 3 | 0 | 3
Infusion site pain (General disorders) | 0 | 1 | 3 | 1 | 7
Malaise (General disorders) | 0 | 0 | 4 | 2 | 5
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 4 | 0 | 20
Pain (General disorders) | 0 | 1 | 0 | 1 | 7
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 4
Pyrexia (General disorders) | 0 | 0 | 7 | 3 | 22
Sluggishness (General disorders) | 0 | 0 | 1 | 0 | 0
Submandibular mass (General disorders) | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 7
Cellulitis (Infections and infestations) | 0 | 0 | 3 | 0 | 3
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 1 | 3
Joint abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Mycobacterium avium complex infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 2 | 9
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 6
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 0 | 8
Tinea pedis (Infections and infestations) | 0 | 1 | 3 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 12 | 2 | 25
Urinary tract infection (Infections and infestations) | 1 | 1 | 2 | 1 | 10
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 8
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 2
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 0 | 13
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood sodium decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood testosterone decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 1 | 0 | 1
Cardiac murmur (Investigations) | 0 | 2 | 0 | 0 | 2
Haematocrit decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 1 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 7
Protein total decreased (Investigations) | 0 | 0 | 1 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 1 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 1 | 4
Weight increased (Investigations) | 0 | 0 | 2 | 1 | 4
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 3
White blood cell count increased (Investigations) | 0 | 0 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 13
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 7
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 6
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 5 | 0 | 15
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5 | 1 | 18
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 1 | 10
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 0 | 12
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 9
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 6
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 5
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 3 | 14
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 5 | 0 | 14
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 4
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 6 | 4 | 26
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 2
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 4 | 0 | 6
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 3
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1
Anger (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 1 | 11
Depression (Psychiatric disorders) | 0 | 1 | 1 | 1 | 5
Insomnia (Psychiatric disorders) | 2 | 2 | 5 | 3 | 29
Irritability (Psychiatric disorders) | 1 | 0 | 2 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 2 | 25
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 5 | 2 | 25
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 2 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 7
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 6
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 3
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 3
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 7
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 1 | 13
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2
Hypertension (Vascular disorders) | 1 | 0 | 2 | 2 | 16
Hypotension (Vascular disorders) | 0 | 0 | 2 | 0 | 3
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.